CLINICAL TRIAL: NCT04213183
Title: Screening and Identifying Hepatobiliary Diseases Via Deep Learning Using Ocular Images
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Huadu Hospital of Southern Medical University (Unknown); Aikang Health Care (Unknown)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: AEHD-2019
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Ophthalmology; Artificial Intelligence; Hepatobiliary Disease
Keywords: Hepatobiliary Disease; Artificial Intelligence; Eye Images
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- development dataset 01: Slit-lamp and retinal fundus images collected from Department of Hepatobiliary Surgery of the Third Affiliated Hospital of Sun Yat-sen University.
  Interventions: Diagnostic Test: Hepatobiliary Disorders
- development dataset 02: Slit-lamp and retinal fundus images collected from Affiliated Huadu Hospital of Southern Medical University.
  Interventions: Diagnostic Test: Hepatobiliary Disorders
- development dataset 03: Slit-lamp and retinal fundus images collected from Nantian Medical Centre of Aikang Health Care.
  Interventions: Diagnostic Test: Hepatobiliary Disorders
- test dataset 01: Slit-lamp and retinal fundus images collected from Department of Infectious Diseases, Third Affiliated Hospital of Sun Yat-sen University.
  Interventions: Diagnostic Test: Hepatobiliary Disorders
- test dataset 02: Slit-lamp and retinal fundus images collected from Huanshidong Medical Centre of Aikang Health Care.
  Interventions: Diagnostic Test: Hepatobiliary Disorders

INTERVENTIONS:
Diagnostic Test: Hepatobiliary Disorders — The training dataset was used to train the deep learning model, which was validated and tested by the other two datasets.

SUMMARY:
Artificial Intelligence may provide insight into exploring the potential covert association behind and reveal some early ocular architecture changes in individuals with hepatobiliary disorders. We conducted a pioneer work to explore the association between the eye and liver via deep learning, to develop and evaluate different deep learning models to predict the hepatobiliary disease by using ocular images.

ELIGIBILITY:
Inclusion Criteria:

* The quality of fundus and slit-lamp images should clinical acceptable.
* More than 90% of the fundus image area including four main regions (optic disk, macular, upper and lower retinal vessel archs) are easy to read and discriminate.
* More than 90% of the slit-lamp image area including three main regions (sclera, pupil, and lens) are easy to read and discriminate.

Exclusion Criteria:

* Images with light leakage (>10% of the area), spots from lens flares or stains, and overexposure were excluded from further analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Slit-lamp and retinal fundus images collected from Department of Infectious Diseases, Third Affiliated Hospital of Sun Yat-sen University, Department of Infectious Diseases, Third Affiliated Hospital of Sun Yat-sen University, Affiliated Huadu Hospital of Southern Medical University, Nantian Medical Centre of Aikang Health Care, and Huanshidong Medical Centre of Aikang Health Care.
Sampling Method: Probability Sample
Enrollment: 1789 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
area under the receiver operating characteristic curve of the deep learning system | baseline
  The investigators will calculate the area under the receiver operating characteristic curve of deep learning system and compare this index between deep learning system and human doctors

SECONDARY OUTCOMES:
sensitivity and specificity of the deep learning system | baseline
  The investigators will calculate the sensitivity and specifity of deep learning system and compare this index between deep learning system and human doctors

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No